CLINICAL TRIAL: NCT02005640
Title: Transcatheter Heart Valve (THV) Sizing and Leakage After Transcatheter Aortic Valve Implantation (TAVI) Before and After Establishing Routine Preprocedure Multi Slice Computerized Tomography (MSCT) Aortic Assessment. A Retrospective Registry Study
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Lars Romer Krusell, MD, Aarhus University Hospital Skejby
Other Study IDs: MSCT-TAVI 1
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MSCT-based prothesis sizing
- Echocardiographic-based prothesis sizing

SUMMARY:
The objective of this study is to evaluate the effect of annular sizing strategy (MDCT versus TEE) in transcatheter aortic valve implantation on the prevalence and severity of paravalvular regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with a THV at Aarhus University Hospital

Exclusion Criteria:

* Learning curve patients (the first 40 patients implanted with a THV device at Aarhus University Hospital, Skejby).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary analysis will be done in patients with a successful THV implantation and availability of high quality echocardiographic assessment and in the post routing MSCT group on the availability of a high quality MSCT scan.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2011-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Rate of no/ mild paravalvular leakage before and after introduction of routing preoperative MSCT | 1 week to 3 months post-TAVI
MSCT vs. echocardiographic aortic valve sizing before TAVI | time of TAVI
THV size before and after introduction of routing preoperative MSCT | time of TAVI

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology and Cardiothoracic Surgery, Aarhus University Hospital, Aarhus N, Denmark